CLINICAL TRIAL: NCT02096328
Title: A Phase II, Open-label, Multi-center Study to Assess Pharmacokinetics (PK), Safety and Efficacy of POL7080 Co-administered With Standard of Care (SoC) Treatment in Patients With Ventilator- Associated Pneumonia (VAP) Due to Suspected or Documented Pseudomonas Aeruginosa Infection.
Brief Title: Pharmacokinetics, Safety and Efficacy of POL7080 in Patients With Ventilator Associated Pseudomonas Aeruginosa Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POL7080-003
Record Dates: First submitted 2014-03-18; First posted 2014-03-26 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2016-06

CONDITIONS: Ventilator Associated Pneumonia; Lower Respiratory Infection
Keywords: Ventilator Associated Pneumonia (VAP); Lower respiratory infection; POL7080; Pseudomonas aeruginosa; Nosocomial pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pseudomonas Infections; Healthcare-Associated Pneumonia | interventions — murepavadin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- POL7080, Anti-pseudomonal antibiotics (Experimental): POL7080 daily co-administered with standard of care treatment
  Interventions: Drug: POL7080

INTERVENTIONS:
Drug: POL7080 — Intravenous infusion

SUMMARY:
To investigate the pharmacokinetic characteristics of POL7080 co-administered with SoC during 10 to 14 days of treatment in VAP patients due to suspected or documented Pseudomonas aeruginosa infection

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years of age diagnosed with VAP , i.e., pneumonia that arises more than 96 hours after endotracheal intubation documented or suspected to be due to Pseudomonas aeruginosa
2. Respiratory specimen suitable for culture and Gram stain collected before starting the treatment
3. Written Informed consent from the patient's legally acceptable representative or a relative

Exclusion Criteria:

1. Patients with known hypersensitivity to fluoroquinolones, carbapenems, cephalosporin, penicillin (beta-lactam antibiotics) or aminoglycoside antibiotics (i.e. all available SoC antibiotics); patients with a clinically significant history of drug allergies and history of anaphylactic reaction and patients with active allergic conditions at the time of screening
2. Known or suspected pulmonary conditions which are likely to interfere with the therapeutic response or might have additional impact on pharmacokinetics
3. Patients with Acute Physiology and Chronic Health Evaluation II (APACHE II) score >25
4. Presence of septic shock at the time of evaluation for study entry
5. History of lung transplant
6. Patients with known HIV infection with CD4+ (cluster of differentiation 4) cell count < 200/mm3
7. Concomitant morbidity of such severity that the patient is likely to die or present with serious medical conditions within 7 days of study entry
8. Patients with impaired renal function
9. Patients who are currently enrolled in, or have not yet completed at least 30 days since ending another investigational device or drug trial or are receiving other investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To measure the plasma concentrations of POL7080 | Day 3 and Day 6
  PK profile of POL7080 will be determined on Day 3 and Day 6.

SECONDARY OUTCOMES:
Adverse Events | Daily assessment up to 34 days from informed consent.
  Number of adverse events reported by the patients or observed by the investigator will be recorded. Onset, end date, severity, causal relationship, outcome and measures taken will be summarized. Death, discontinuations and serious adverse events will be listed and narrative summaries will be provided.
Laboratory abnormalities | Day 4, Day 6, Day 10, Day 15, Day 24 and Day 34
  The number and severity of blood chemistry and hematology abnormal findings will be summarized descriptively and compared to baseline. Clinically significant values/outliers will be listed and commented.

OTHER OUTCOMES:
Clinical cure | Day 4, Day 6, Day 10, Day 15, Day 24 and Day 34
  Clinical cure will be measured based on clinical signs and symptoms and radiological findings.
Reduction in bacterial count | Day 4, Day 6, Day 10, Day 15, Day 24 and Day 34
  Reduction in CFU/mL (colony forming unit /mL) of Pseudomonas aeruginosa in the daily quantitative cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Torres, MD PhD, Principal Investigator — Hospital Clinic, Barcelona, SPAIN; Evangelos Giamarellos-Bourboulis, MD PhD, Principal Investigator — ATTIKON University Hospital, Athens, GREECE
Locations (10):
- Greece (4):
  - ATTIKON University Hospital, Athens
  - Hospital EVANGELISMOS, Athens
  - Hospital KORGIALENIO-BENAKIO E.E.S, Athens
  - SOTIRA Pulmonary Clinic, Athens
- Spain (6):
  - Hospital Bellvitge, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Del Mar, Barcelona
  - Hospital Clinic San Carlos, Madrid
  - Hospital Joan XXIII, Tarragona
  - Hospital La Fe, Valencia